CLINICAL TRIAL: NCT03606577
Title: An Intensive Program With Quadruplet Induction and Consolidation Plus Tandem Autologous Stem Cell Transplantation in Newly Diagnosed High Risk Multiple Myeloma Patients: a Phase II Study of the Intergroupe Francophone du Myélome "IFM 2018-04"
Brief Title: An Intensive Program With Quadruplet Induction and Consolidation Plus Tandem Autologous Stem Cell Transplantation in Newly Diagnosed High Risk Multiple Myeloma Patients
Acronym: IFM 2018-04
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC18_0206
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Newly Diagnosed; High Risk; Revlimid; Carfilzomib; Daratumumab; Dexaméthasone
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: One group of subjects who must have documented Multiple Myeloma High Risk satisfying the CRAB and measurable disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carfilzomib, Daratumumab, Lenalidomide and Dexaméthasone (Experimental)
  Interventions: Drug: Carfilzomib; Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Induction 6 cycles 20/36 mg/m² on days 1, 2, 8, 9, 15, 16 (20 mg/m² on D1 and 2 cycle 1 only) Consolidation 4 cycles Carfilzomib 20 or 36 mg/m² on days 1, 2, 8, 9, 15, 16 (20 mg/m² on D1 and 2 first cycle only)
Drug: Daratumumab — induction: 6 cycles Daratumumab 8/16mg/kg IV on Days 1, 8, 15, 22 for the first two cycle 2 and on days 1 and 15 for cycles 3 to 6. (8mg/kg on D1 & D2 cycle 1 only) Consolidation: daratumumab 4 cycles 16mg/kg IV Day 1, Day 15 Maintenance Daratumumab 16mg/kg IV once every 8 weeks for 2 years (or until documented disease progression)
Drug: Lenalidomide — induction: 6 cycles Lenalidomide 25 mg/day from day 1 to day 21 Consolidation: 4 cycles 15 mg/day from Day 1 to Day 21 (first cycle ) 25 mg/day from Day 1 to Day 21 (in the following cycle) Maintenance therapy 10mg/day, Day 1 to 21, for 2 years (or until documented disease progression)
Drug: Dexamethasone — induction 6 cycles 20 mg/day on days 1-2, 8-9, 15-16 and 22-23 Consolidation 4 cycles 40 mg/Day on Days 1, 8, 15 and 22

SUMMARY:
According to international guidelines, upfront therapy for transplant eligible myeloma patients should include triplet induction containing proteasome inhibitor and immunomodulatory agent, autologous stem cell transplant, PI+Imid based triplet consolidation and lenalidomide maintenance. Despite this approach, virtually all MM patients experience disease relapse, especially those with High Risk disease defined by adverse cytogenetic abnormalities (i.e. del(17p), or t(14;16) or t(4;14)) detected by FISH and/or SNP arrays. Indeed, HR myeloma is associated with poorer progression free survival and overall survival and frontline therapy should therefore be improved for this subset of HR patients. The primary objective of this prospective multicenter, open label, interventional phase 2 trial is to evaluate the feasibility of an intensive program including quadruplet induction and consolidation, tandem autologous stem cell transplantation and maintenance in newly diagnosed multiple myeloma patients presenting with HR cytogenetic. Quadruplet induction and consolidation include carfilzomib, lenalidomide, dexamethasone and daratumumab. Maintenance will include lenalidomide and daratumumab. Secondary objectives will include efficacy parameters (i.e. response rate, minimal residual disease, safety, progression free survival, overall survival).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 years of age or older, younger than 66 years (< 66 years)
2. Voluntary written informed consent must be given before performance of any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
3. Subject must have documented multiple myeloma satisfying the Diagnostic criteria for symptomatic Myelome Multiple and measurable disease as defined by:

   * Monoclonal plasma cells in the bone marrow ≥ 10% or presence of a biopsy proven plasmacytoma AND any one or more of the following myeloma defining events:

     * Hypercalcemia: serum calcium > 0.25 mmol/L higher than ULN or > 2.75 mmol/L
     * Renal insufficiency: creatinine clearance < 40mL/min or serum creatinine > 177 μmol/L
     * Anemia: hemoglobin > 2 g/dL below the lower limit of normal or hemoglobin < 10 g/dL
     * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT or PET-CT Or in a patient with indolent myeloma
     * Clonal bone marrow plasma cell percentage ≥ 60%
     * Involved: uninvolved serum free light chain ratio ≥ 100
     * Superior 1 focal lesion on MRI studies
   * Measurable disease as defined by the following:

   M-component ≥ 5g/l, and/or urine M-component ≥ 200 mg/24h and/or serum Free Light Chain ≥ 100 mg/l.
4. Newly diagnosed subjects eligible for high dose therapy and autologous stem cell transplantation
5. Subject must have high risk disease according to FISH analysis: del(17p), or t(14;16) or t(4;14). The FISH-positivity cut-off value for defining the presence of del(17p) in this study is 50%
6. Karnofsky performance status score ≥ 50%
7. Women of childbearing potential must have a negative serum or urine pregnancy test within 10 to 14 days prior to therapy and repeated within 24 hours before starting study drug. They must commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control used at the same time, beginning at least 4 weeks before initiation of lenalidomide treatment and continuing for at least 30 days after the last dose of Lenalidomide. Women must also agree to notify pregnancy or doubt upon pregnancy during the study.
8. Men must agree to not father a child and agree to use a latex condom during therapy and for 4 weeks after the last dose of study drug, even if they have had a successful vasectomy, if their partner is of childbearing potential.
9. Subject must have pretreatment clinical laboratory values meeting the following criteria during the Screening Phase (Lab tests should be repeated if done more than 15 days before C1D1):

   1. Hemoglobin ≥ 7.5 g/dL. Prior red blood cell transfusion or recombinant human erythropoietin use is permitted;
   2. Absolute neutrophil count ≥ 1.0 Giga/l (GCSF use is permitted);
   3. ASAT ≤ 3 x ULN;
   4. ALAT ≤ 3 x ULN;
   5. Total bilirubin ≤ 3 x ULN (except in subjects with congenital bilirubinemia, such as Gilbert syndrome, direct bilirubin ≤ 1.5 x ULN);
   6. Calculated creatinine clearance ≥ 40 mL/min/1.73 m² ;
   7. Corrected serum calcium ≤ 14 mg/dL; or free ionized calcium ≤6.5 mg/dL;
   8. Platelet count ≥ 50 Giga/l for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; otherwise platelet count > 50 Giga/l (transfusions are not permitted to achieve this minimum platelet count).
10. Affiliation with French social security system or beneficiary from such system

Exclusion Criteria:

1. Subjects must not have been treated previously with any systemic therapy for multiple myeloma. Prior treatment with corticosteroids or radiation therapy does not disqualify the subject (the maximum dose of corticosteroids should not exceed the equivalent of 160 mg of dexamethasone in a 2-week period). Two weeks must have elapsed since the date of the last radiotherapy treatment. Enrolment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 2 weeks have elapsed since the last date of therapy
2. Subject has received daratumumab or other anti-CD38 therapies previously
3. Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, or solitary plasmacytoma.
4. Subject has a diagnosis of Waldenström's macroglobulinemia, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
5. Subject has had plasmapheresis within 28 days of C1D1.
6. Subject is exhibiting clinical signs of meningeal involvement of multiple myeloma.
7. Myocardial infarction within 6 months prior to enrolment according to NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
8. Uncontrolled hypertension
9. Subjects with known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume (FEV1) in 1 second < 50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 < 50% of predicted normal.
10. Subjects with a history of moderate or severe persistent asthma within the past 2 years, or with uncontrolled asthma of any classification at the time of screening (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
11. Subject has plasma cell leukemia (according to WHO criterion: ≥ 20% of cells in the peripheral blood with an absolute plasma cell count of more than 2 × 10^9/L) or polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes syndrome.
12. Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (as clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (as rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, fosphenytoin phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment.
13. Known intolerance to steroid therapy
14. History of hypersensitivity to any of the study medications, their analogues, or excipients in the various formulations, or to study-required co medication
15. Subject has had major surgery within 2 weeks before the first dose of study treatment or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study. Kyphoplasty or Vertebroplasty are not considered major surgery.
16. Clinically relevant active infection or serious co-morbid medical conditions
17. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer free of disease since 5 years.
18. Female subject who is pregnant or breast-feeding + male and female refusing birth control conditions
19. Serious medical or psychiatric illness likely to interfere with participation in study
20. Uncontrolled diabetes mellitus
21. Known HIV infection; Known active hepatitis B or C viral infection; or other ongoing uncontrolled infection
22. Incidence of gastrointestinal disease that may significantly after the absorption of oral drugs
23. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment
24. Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-02-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients receiving the second Autologous Stem Cell Transplant | 15 months

SECONDARY OUTCOMES:
Number of adverse events | 48 months
Number of responses | 48 months
Number of MRD | 48 months
Number of death | 84 months
Percentage of time to progression | 84 months
Number of patients having survival without progress | 84 months
Percentage duration of response | 84 months
Number of cells collected | 168 days
percentage of value of biological prognostic factors | 48 months

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de Nantes, Nantes, Pays de la Loire Region
  - CHU Caen, Caen
  - CHRU Dijon, Dijon
  - CHRU - Hôpital A.Michallon, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHRU - Hôpital Claude Huriez, Lille
  - CH de Lyon Sud, Lyon
  - CHRU Hôpital du Haut Lévêque, Pessac
  - CHRU - Hôpital de Pontchaillou, Rennes
  - CHU Toulouse, Toulouse
  - CHRU Bretonneau, Tours
  - CHRU - Hôpitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Touzeau C, Perrot A, Hulin C, Manier S, Macro M, Chretien ML, Karlin L, Escoffre M, Jacquet C, Tiab M, Leleu X, Avet-Loiseau H, Jobert A, Planche L, Corre J, Moreau P. Daratumumab, carfilzomib, lenalidomide, and dexamethasone with tandem transplant for high-risk newly diagnosed myeloma. Blood. 2024 May 16;143(20):2029-2036. doi: 10.1182/blood.2023023597. PMID 38394666
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481